CLINICAL TRIAL: NCT02944773
Title: Assessment of Facilitated Tucking During the Procedure of Daily Weight on the Level of Stress in Preterm Infants
Acronym: UTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IIBSP-EST-2015-97
Record Dates: First submitted 2016-10-10; First posted 2016-10-26 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2017-12

CONDITIONS: Stress
Keywords: newborn; facilitated tucking; position; weight; stress
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- facilitated tucking device (FTD) (Experimental): 20 infants use a FTD in the procedure of daily weight
  Interventions: Procedure: Facilitated tucking device
- without FTD (No Intervention): 20 infants use not a FTD in the procedure of daily weight

INTERVENTIONS:
Procedure: Facilitated tucking device — 20 newborns are using a facilitated tucking device weight during the procedure to assess the level of stress
  Arms: facilitated tucking device (FTD)

SUMMARY:
Randomized crossover clinical trial in which is intended to assess the effect of facilitated tucking of premature infants during daily weight. Heart rate, respiratory rate and neo-scale stress (ALPS-Neo) be observed before, during and one hour after the weight, and compared with normal practice, without facilitated tucking device.

DETAILED DESCRIPTION:
Population(n): 20 newborn When a patient is a possible candidate, consent will be asked their parents. After obtaining informed consent signed by parents, it will be assigned a random group (G1, G2). In the G1, the first weight without facilitated tucking device and the next day with facilitated tucking device will be held. G2 will be done in reverse.

Handling pre phase (T0): at least 20 minutes before vitals heart rate and respiratory rate are taken in five times.

handling phase (T1): 1. the facilitated tucking device is placed. 2. will wait five minutes and weight will be held in the incubator;at the time of leaving it in the incubator the same constants are taken.

post handling phase (T2): the same constants are taken one hour after such manipulation.

ELIGIBILITY:
Inclusion Criteria:

* ≤1500 grams newborns
* a week of life about

Exclusion Criteria:

* Surgery
* Hemodynamic instability requiring vasoactive drugs
* Sedation
* Phototherapy at the time of the procedure
* Congenital anomalies.

Ages: 5 Days to 9 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Heart rate and breathing rate will be decreased compared to baseline measurement. | one year
  Heart rate (beats / minute)and respiratory rate will decrease significantly during facilitated tucking weight.

SECONDARY OUTCOMES:
Behavioral signs | one year
  ALPS-Neo scale will decreased significantly during facilitated tucking weight. Evaluate the behaviors: facial expression, respiratory pattern, tone of limbs, activity of hands and feet, and level of activity collected on the scale ALPS-Neo during weight, and compare them with facilitated tucking weight

CONTACTS AND LOCATIONS:
Overall Officials: silvia Vicente Pérez, Principal Investigator — Fundació de Gestió Sanitària de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Silvia Vicente Pérez, Castelldefels, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
october 2017